CLINICAL TRIAL: NCT07296146
Title: Effect of Probiotic Supplementation on Resistant Anaemia to Erythropoietin in Chronic Kidney Disease Patients.
Brief Title: Probiotics Against Erythropoietin Resistance in Chronic Kidney Disease Patients.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Eman Said Sawan, Lecturer, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 121-2025
Record Dates: First submitted 2025-11-19; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Anaemia; Chronic Kidney Disease; Regular Hemodialysis
Keywords: Probiotic; erythropoietin; resistant anaemia; chronic kidney disease patients
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Erythropoietin; Probiotics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPO + Probiotic (Active Comparator): EPO (4000 IU) + Probiotic (Lactobacillus acidophilus, 5 billion)
  Interventions: Drug: Erythropoietin + Probiotic
- EPO (Active Comparator): Erythropoietin (Epoetin 4000 IU)
  Interventions: Drug: EPO

INTERVENTIONS:
Drug: Erythropoietin + Probiotic — Anaemic chronic kidney disease patients on regular hemodialysis treated with Erythropoietin + Probiotic
  Arms: EPO + Probiotic
Drug: EPO — Anaemic chronic kidney disease patients on regular hemodialysis treated with Erythropoietin
  Arms: EPO

SUMMARY:
The goal of this clinical trial is to assess whether probiotic supplementation can improve the hematological response of CKD patients to erythropoietin therapy and prevent or reduce erythropoietin resistance. The main questions it aims to answer are:

Can probiotic be used as an adjuvant strategy in anemia management and increasing ESA responsiveness in CKD? What medical problems do participants have when taking probiotic? Researchers will compare Erythropoietin only with Erythropoietin + Probiotic to see if Probiotic aids in treating anaemic chronic kidney disease patients.

Participants will:

Take Erythropoietin + Probiotic or Probiotic only every day for 3 months Visit the clinic once every 4 weeks for checkups and tests Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with end stage renal disease for more than 3 months on regular hemodialysis (GFR less than 15 ml/min/m2
* Receiving stable doses of erythropoietin therapy
* Able and willing to provide informed consent

Exclusion Criteria:

* Recent probiotic, antibiotic, or immunosuppressive therapy
* Microcytic hypochromic anemia.
* Patients with hyperparathyroidism
* Recent or planned kidney transplantation Gastrointestinal disorders (active IBD, cancer)
* Pregnancy or lactation
* Severe comorbidities (e.g., active infection, malignancies)
* Cognitive or physical inability to comply with protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
- Hemoglobin concentration | at baseline, and 3-months postintervention
  - Hemoglobin concentration (g/dL)at 2 weeks, and 3-months postoperatively
- Erythropoietin resistance index (ERI) | at baseline, and 3-months postintervention
  - ERI = (ESA dose per week) / (body weight) / (hemoglobin level).

SECONDARY OUTCOMES:
C-reactive protein | at baseline, and 3-months postintervention
  mg/dl
serum urea | at baseline, and 3-months postintervention
  mg/dl

IPD SHARING:
Plan to Share IPD: No